CLINICAL TRIAL: NCT00018148
Title: Combined Nortriptyline and Transdermal Nicotine for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Prochazka, Allan - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADRD-006-97F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Smoking
Keywords: smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nortriptyline; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Transdermal nicotine plus nortriptyline
  Interventions: Drug: nortriptyline
- 2 (Active Comparator): Transdermal nicotine plus placebo
  Interventions: Drug: transdermal nicotine

INTERVENTIONS:
Drug: nortriptyline — Dose titrated to 75 mg daily as tolerated combined with transdermal nicotine 21 mg
  Arms: 1
Drug: transdermal nicotine — Transdermal nicotine 21 mg, titrated down plus placebo
  Arms: 2

SUMMARY:
Treatment of smokers with a tricyclic antidepressant, nortriptyline, can reduce tobacco withdrawal symptoms and increases long term cessation rates when combined with transdermal nicotine and a behavioral cessation programs. The study is a placebo-controlled, randomized, parallel group trial in which smokers aged 18-70 will be subject to the combination of oral and patch treatments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70,
* smoking > 10 cigarettes per day,
* no current major depression,
* no concurrent psychiatric medications

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 1998-04; Primary Completion 2002-12 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Validated smoking cessation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan V. Prochazka, MD MSc, Principal Investigator — VA Eastern Colorado Health Care System, Denver
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

REFERENCES:
- [Result] Prochazka AV, Kick S, Steinbrunn C, Miyoshi T, Fryer GE. A randomized trial of nortriptyline combined with transdermal nicotine for smoking cessation. Arch Intern Med. 2004 Nov 8;164(20):2229-33. doi: 10.1001/archinte.164.20.2229. PMID 15534159
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961